CLINICAL TRIAL: NCT01096316
Title: Reducing Disparities and Improving Care for Depression in OB-GYN Clinics: Depression Attention for Women Now (The DAWN Study)
Brief Title: Depression Attention for Women Now (The DAWN Study)
Acronym: DAWN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jurgen Unutzer, Professor and Chair, Psychiatry & Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37061-G; 1R01MH085668 (NIH)
Record Dates: First submitted 2010-03-25; First posted 2010-03-31 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Depressive Disorder
Keywords: mood disorders; depressive disorder; women; depression
MeSH Terms: conditions — Depressive Disorder; Mood Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The intervention will integrate care between a depression care manager, consulting study team (psychiatry, psychology, OB-GYN researchers) and OB-GYN clinic providers. The 3-part intervention includes:
  * enhanced education of patients and providers
  * engagement of patients
  * depression care management with patient choice of initial antidepressant medication or Problem-Solving Treatment-Primary Care and behavioral activation.
  Interventions: Behavioral: Depression Care Management
- Usual Care (No Intervention): Patients randomized to Usual Care Arm will be informed of their diagnosis and encouraged to inform her OB-GYN provider about her depression diagnosis. Patients will be encouraged to proceed with care using any primary care or specialty services normally available to them inside/outside their OB-GYN clinic. All treatment decision for Usual Care Arm patients are left to the OB-GN provider.

INTERVENTIONS:
Behavioral: Depression Care Management — The intervention is conducted by a social worker who has the role of a Depression Care Manager (DCM). First, a unique engagement session develops rapport with the DCM, providing education and identifying health concerns. DCM meets in-person and/or by phone every 1-2 weeks for 12 weeks, then monthly for the rest of the 12-month intervention. Patients choose either medication or Problem-Solving Treatment-Primary Care therapy. Depressive symptoms are assessed at each visit with the PHQ-9, as well as response to medications or to PST, with a total of 8 PST-PC sessions. Patients with inadequate response after 8 weeks to the first choice will switch or combine treatments. Providers are given extensive feedback about the patient's health care concerns.
  Other Names: Study Intervention
  Arms: Intervention

SUMMARY:
Major depressive disorder (MDD) is a common disabling illness that disproportionately affects women, with prevalence rates two times those of men. In addition to suffering, MDD has been shown to have a marked effect on social and vocational functioning, with increased disability, lost productivity, and excess mortality. Women with MDD have an increased prevalence of comorbid anxiety disorders and medical conditions.

Our model of care utilizes a social worker as a depression care manager (DCM) to support both patients and physicians in optimizing care in the OB-GYN clinical setting. This intervention will be compared to usual care for depression.

DETAILED DESCRIPTION:
A large number of women receive their routine care in OB-GYN clinics, including a disproportionate percentage of low-income and minority women. For many of these women, OG-GYNs are the only provider they see on a regular basis. OB-GYNs take care of women across their lifespan, addressing gynecologic, health care maintenance, pregnancy and primary care concerns in their everyday practices. There are multiple aspects of OG-GYN care that are uniquely suited for detection and treatment of depression, but there are also significant barriers to such care that must be addressed.

In this randomized controlled trial, we are testing this depression care management program for women attending two OB-GYN clinics in the University of Washington health care system. Our research aims to test the hypothesis that a depression care management intervention, integrated into the OB-GYN clinic setting, will improve treatment outcomes for depression, functional outcomes, and satisfaction with depression care. The results of our research will greatly impact clinical care by satisfying an unmet need for effective depression services for women seen in OB-GYN clinical settings.

The study compares a depression care management intervention, delivered by a depression care manager, to usual care for depression in the clinics. The primary aims of the study are to evaluate, compared to usual care, a depression intervention consisting of enhanced education, engagement, and depression care management (with a choice of antidepressant medication monitoring and/or provision of brief psychotherapy).

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 score ≥10 for Major Depressive Disorder (with 1 cardinal symptom) and/or ≥10 for Dysthymia (with 1 cardinal symptom)
* MINI confirmation of PHQ-9 diagnoses
* Access to a telephone
* English-speaking

Exclusion Criteria:

* High suicide risk (PHQ-9 response)
* ≥2 prior suicide attempts
* Lifetime history of schizophrenia or bipolar disorder (MINI response)
* Substance abuse/dependence within the previous 3 months (CAGE-AID)
* Current severe intimate partner violence
* Currently seeing a psychiatrist

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2009-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Unutzer, MD, MPH, MA, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Women's Clinic at Harborview Medical Center, Seattle, Washington
  - Women's Health Care Center at University of Washington Medical Center (Roosevelt Clinic), Seattle, Washington

REFERENCES:
- [Result] Melville JL, Reed SD, Russo J, Croicu CA, Ludman E, LaRocco-Cockburn A, Katon W. Improving care for depression in obstetrics and gynecology: a randomized controlled trial. Obstet Gynecol. 2014 Jun;123(6):1237-1246. doi: 10.1097/AOG.0000000000000231. PMID 24807320
- [Result] Cerimele JM, Vanderlip ER, Croicu CA, Melville JL, Russo J, Reed SD, Katon W. Presenting symptoms of women with depression in an obstetrics and gynecology setting. Obstet Gynecol. 2013 Aug;122(2 Pt 1):313-318. doi: 10.1097/AOG.0b013e31829999ee. PMID 23969800
- [Result] LaRocco-Cockburn A, Reed SD, Melville J, Croicu C, Russo JE, Inspektor M, Edmondson E, Katon W. Improving depression treatment for women: integrating a collaborative care depression intervention into OB-GYN care. Contemp Clin Trials. 2013 Nov;36(2):362-70. doi: 10.1016/j.cct.2013.08.001. Epub 2013 Aug 9. PMID 23939510

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: The intervention will integrate care between a depression care manager, consulting study team (psychiatry, psychology, OB-GYN researchers) and OB-GYN clinic providers. The 3-part intervention includes:
  * enhanced education of patients and providers
  * engagement of patients
  * depression care management with patient choice of initial antidepressant medication or Problem-Solving Treatment-Primary Care and behavioral activation.
  Depression Care Management: The intervention is conducted by a social worker who has the role of a Depression Care Manager (DCM). First, a unique engagement session develops rapport with the DCM, providing education and identifying health concerns. DCM meets in-person and/or by phone every 1-2 weeks for 12 weeks, then monthly for the rest of the 12-month intervention. Patients choose either medication or Problem-Solving Treatment-Primary Care therapy. Depressive symptoms are assessed at each visit with the PHQ-9, as well as response to medications or to PST,
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 102 | 103
Completed | 87 | 94
Not Completed | 15 | 9
Not completed — Lost to Follow-up | 15 | 9

BASELINE CHARACTERISTICS:
Population: Baseline data from the intervention arms were examined for statistically significant differences using t tests, chi squares and logistic regression analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 102 | 103 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.47 (12.11) | 38.59 (12.10) | 39.02 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 103 | 205
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Depression Treatment Outcome
Description: Impact of the intervention on depression treatment outcomes, including change in depressive symptoms and treatment response. In particular, the depression scale from the Hopkins Symptom Checklist 20 (SCL-20) was used to assess depression severity at the assessments. The SCL-20 ranges from 0 (no depression) to 4 (severe depression),
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 102 | 103
units on a scale | 0.96 (0.65) | 1.33 (0.75)

2. Primary Outcome: Functional Outcome
Description: Impact of the intervention on functional outcomes of patients. Functional impairment was measured using the Sheehan Disability Scale. The Sheehan disability scale is the average of 3 items assessing impairment in social, work and family responsibilities. Each item is rated 0 (no impairment) to 10 (totally impaired) and the 3 ratings are averaged for the Sheehan disability scale reported below.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 102 | 103
units on a scale | 3.69 (2.70) | 4.03 (2.70)

3. Secondary Outcome: Quality of Depression Care Indicators
Description: Intervention impact on quality of depression care indicators and satisfaction with depression care. Number of participants receiving 4 or more mental health visits are reported. Receiving 4 or more mental health visits has previously been used in depression randomized control trials as a measure of the quality of depression treatment received by a patient
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 102 | 103
participants | 67 | 28

4. Secondary Outcome: Potential Facilitators and Barriers to Sustainability
Description: Providers' and administrators' perceived barriers and facilitators to continue providing the intervention after study end.
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Intervention: The intervention will integrate care between a depression care manager(DCM), consulting study team (psychiatry OB-GYN physician) and OB-GYN clinic providers.
  Depression Care Management: The intervention is conducted by a social worker who has the role of a Depression Care Manager (DCM). The DCM in a unique engagement session develops rapport with the DCM, providing education and identifying health concerns. DCM meets in-person and/or by phone every 1-2 weeks for 12 weeks, then monthly for the 12-month intervention. Patients choose either medication or Problem-Solving Treatment. Depressive symptoms are assessed at each visit with the PHQ-9. Patients with inadequate response after 4 to 8 weeks to the first choice will switch or combine treatments. DCMs partcipate in weekly caseload review with a psychiatrist and Ob-Gyn physician who make treatment recommendations that the DCM then communicates to the patient's own Ob-Gyn physician who writes all prescriptions.
Arm/Group | Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 1/102 | 1/103
Other Adverse Events (participants affected / at risk) | 0/102 | 0/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=102) | Usual Care (N=103)
Psychiatric ER visits or hospitalization (Psychiatric disorders) | 1 (1) | 1 (1) — We assessed at each objective follow-up all psychiatric emergency room visits and psychiatric hospitalizations. These were also spontaneously sent to us via EMR if the ER visit or hospitalization occurred in the University hospitals

LIMITATIONS AND CAVEATS:
Patients were recruited from university-affiliated OB/GYN clinics, which potentially limits generalizability to other OB/GYN populations; non-English speaking women were not included; and antidepressant adherence was based on self-report data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes